CLINICAL TRIAL: NCT02145390
Title: A Phase II Study of Chemoradiation for Bladder Preservation in Patients With Muscle Invasive Bladder Carcinoma After Complete Response to Neoadjuvant Chemotherapy
Brief Title: Chemoradiation for Bladder Preservation After Complete Response to Neoadjuvant Chemotherapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator Decision - Insufficient Accrual
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Adrian Ishkanian, Assistant Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20130896
Record Dates: First submitted 2014-05-20; First posted 2014-05-22 (Estimated); Results first posted 2018-08-28 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Bladder Cancer; Bladder Carcinoma; Transition Cell Cancer; Muscle Invasive Bladder Carcinoma
Keywords: Bladder Cancer; Bladder Carcinoma; Transition Cell Cancer; TCC; Muscle Invasive Bladder Carcinoma
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Cystoscopy; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TURBT, NAC and Chemoradiation (Experimental): * Transurethral Resection of the Bladder Tumor & Cystoscopy (TURBT);
  * Neoadjuvant Chemotherapy (NAC), per standard of care: Cisplatin and Gemcitabine therapy, within 8 weeks following the TURBT and cystoscopic evaluation;
  * For subjects with complete response (CR): Chemoradiation within 6 weeks after post-neoadjuvant evaluation. Intensity Modulated Radiation Therapy (IMRT/VMAT); Cisplatin therapy per standard of care;
  * For subjects who have pT1 or worse tumor response: Radical Cystectomy, per standard of care, within 12 weeks post-neoadjuvant chemotherapy evaluation;
  * Expanded Prostate Cancer Index Composite Short Form 12 (EPIC SF-12);
  * International Prostate Symptom Score (IPSS).
  Interventions: Procedure: Transurethral Resection of the Bladder Tumor & Cystoscopy; Radiation: Intensity Modulated Radiation Therapy; Behavioral: Expanded Prostate Cancer Index Composite Short Form 12; Behavioral: International Prostate Symptom Score

INTERVENTIONS:
Procedure: Transurethral Resection of the Bladder Tumor & Cystoscopy — TURBT and Cystoscopy will be performed by the participating urologist prior to start of neoadjuvant chemotherapy, per the study protocol:
  * Cystoscopic evaluation
  * Bimanual examination under anesthesia,
  * Transurethral resection of the bladder tumor,
  * Biopsy of the prostatic urethra including both mucosa and stroma using a resection loop.
  Other Names: TURBT
Radiation: Intensity Modulated Radiation Therapy — For subjects with complete response to neoadjuvant chemotherapy. Subjects will receive 25 daily fractions (5 weeks) of radiation therapy for 5 days a week (Monday to Friday) except on weekends or holidays, when remaining fractions will be added to the end of treatment. The overall schema is for IMRT based radiation to the entire bladder, prostate (in men) and the pelvic lymph nodes:
  * Pelvic lymph nodes: 45 Gy in 25 fractions at 1.8 Gy per fraction.
  * Whole bladder and prostate: 50 Gy in 25 fractions at 2.0 Gy per fraction.
  * Tumor boost area: 60-65 Gy in 25 fractions at 2.4-2.6 Gy per day
  * Final boost dose will be determined at the discretion of the treating physician based on normal tissue exposure and volume.
  Other Names: IMRT; VMAT
Behavioral: Expanded Prostate Cancer Index Composite Short Form 12 — Quality of life questionnaire to be administered to subjects at intervals defined by the study protocol.
  Other Names: EPIC SF-12
Behavioral: International Prostate Symptom Score — Quality of life questionnaire to be administered to subjects at intervals defined by the study protocol.
  Other Names: IPSS

SUMMARY:
Bladder preservation in patients with complete response after neoadjuvant chemotherapy will lead to equivalent or superior relapse free rates compared to cystectomy rates from historical controls.

DETAILED DESCRIPTION:
1. Transurethral Resection of the Bladder Tumor (TURBT) and Cystoscopy performed by participating urologist:

   * cystoscopic evaluation
   * bimanual examination under anesthesia,
   * as thorough as possible a transurethral resection (TUR) of the bladder tumor,
   * and a biopsy of the prostatic urethra including both mucosa and stroma using a resection loop.
2. Neoadjuvant Chemotherapy, per standard of care: All patients will receive the neoadjuvant course of chemotherapy. The recommended neoadjuvant chemotherapy regimen consists of Gemcitabine and Cisplatin given on a 21-day cycle.This regimen will begin within 8 weeks following the TURBT and cystoscopic evaluation by the urologic surgeon;
3. Post-Neoadjuvant Evaluation: This evaluation will take place ≤ 6 weeks following the completion of the neoadjuvant chemotherapy. Evaluation will include:

   * urine cytology,
   * cystoscopy,
   * tumor site transurethral biopsy,
   * and bimanual examination after biopsy
   * and biopsy of TURBT site
4. For subjects with complete response to neoadjuvant chemotherapy: Chemoradiation within 6 weeks after post-neoadjuvant evaluation. Intensity Modulated Radiation Therapy (IMRT/VMAT), and concurrent Cisplatin therapy, per standard of care; OR
5. For subjects with pT1 or worse tumor response to neoadjuvant chemotherapy: Radical Cystectomy within 12 weeks after post-neoadjuvant evaluation;
6. Post-Consolidation Endoscopic Evaluations: The first post-treatment evaluation will be 30 days +/- 14 days within the end of chemoradiation, surgery or at progression. Subsequent cystoscopic evaluation will be every three months in the first year, every four months in the second year, and every six months in the third year (all evaluations to occur +/- 14 days). Each evaluation will include serum, plasma, whole blood, urine cytology.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically proven diagnosis of primary carcinoma of the bladder(transitional cell cancer). Must be operable patients with muscularis propria invasion and American Joint Committee on Cancer (AJCC) clinical stages T2-4a, N0 or N+, M0. Patients with prostatic urethra involvement with transitional cell cancer (TCC) are eligible if it is completely resected and the patient has no evidence of stromal invasion of the prostate.
2. Patients must be able to tolerate systemic chemotherapy combined with pelvic radiation therapy and radical cystectomy.
3. Zubrod Performance Status of ≤1.
4. Age ≥18.
5. Complete Blood Count (CBC)/differential obtained no more than 8 weeks prior to enrollment on study, with adequate bone marrow function defined as follows:

   * White Blood Cell (WBC) ≥ 4000/ml
   * Absolute neutrophil count (ANC) ≥1,800 cells/mm
   * Platelets ≥100,000 cells/mm
   * Hemoglobin ≥ 10.0 mg/dl (Note: the use of transfusion or other intervention to achieve this level is acceptable)
6. Serum bilirubin of 2.0mg or less;
7. Serum creatinine of 1.5mg or less; creatinine clearance of 60ml/min or greater no more than 8 weeks prior to enrollment (Note: calculated creatinine clearance is permissible, using Cockcroft-Gault formula. If the creatinine clearance is greater than 60ml/min, then a serum creatinine of up to 1.8mg is allowable at the discretion of the principal investigator.)

   Note: Prechemotherapy laboratory investigations and Eastern Cooperative Oncology Group (ECOG) evaluation must meet inclusion criteria irrespective of where they were drawn, retroactive, prior to cycle 1 of cisplatin/gemcitabine. Inclusion criteria from these initial investigations will be used for evaluation of enrollment eligibility.
8. Patients must be willing and able to provide study-specific informed consent prior to study entry

Exclusion Criteria:

1. Tumor related untreated active hydronephrosis
2. Evidence of distant metastases.
3. Diffuse bladder carcinoma in situ (CIS) not able to be encompassed in a boost radiotherapy volume.
4. Previous systemic chemotherapy (for any cancer) or pelvic radiation therapy
5. A prior or concurrent malignancy of any other site or histology unless the patient has been disease free for greater than or equal to five years except for non-melanoma skin cancer and/or stage T1a prostate cancer or carcinoma in situ of the uterine cervix
6. Patients that are not candidates for radical cystectomy (T4b disease are considered unresectable)
7. Pregnancy or women of childbearing potential [not post-menopausal or permanently sterilized (e.g. tubal occlusion, hysterectomy, bilateral salpingectomy)] and men who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic
8. Severe active co-morbidity:

   * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
   * Transmural myocardial infarction within the last 6 months
   * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
   * Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of enrollment
   * History of hepatic insufficiency resulting in clinical jaundice and/or coagulation defects (Note: laboratory tests for liver function and coagulation parameters are not required for enrollment into this protocol)
   * Known diagnosis of Acquired Immune Deficiency Syndrome (AIDS) based upon current Centers for Disease Control (CDC) definition (Note: HIV testing is not required for enrollment into this protocol). The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive.
   * As determined by the investigator or principal investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-01-05 (Actual); Primary Completion 2017-04-25 (Actual); Study Completion 2017-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian S Ishkanian, MD, Principal Investigator — University of Miami Sylvester Comprehensive Cancer Center
Locations (1):
- University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TURBT, NAC and Chemoradiation
Started | 1
Completed | 0
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | TURBT, NAC and Chemoradiation
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Rate of Failure-Free Survival With Intact Bladder (FFSIB) in Study Participants
Description: Rate of failure free survival with intact bladder (FFSIB) at two years in subjects undergoing bladder preservation. FFSIB is defined by the absence of any failures (locoregional, distant metastasis, and death) and bladder preservation (no radical cystectomy for any causes) after definitive chemoradiation. FFSIB is defined as the time elapsed from the start of neoadjuvant chemotherapy to the date of documented failure events or radical cystectomy. For failure-free patients (without failure events and no radical cystectomy), FFSIB will be censored at the last date of documented failure-free bladder preservation (FFBP) status.
Time Frame: 2 years
Population: A minimum of 35 evaluable participants were required for the analysis of this outcome measure. Fewer than 35 participants were enrolled therefore data were not analyzed.
Arm/Group | TURBT, NAC and Chemoradiation
Number analyzed (Participants) | 0

2. Secondary Outcome: Rate of Failure-Free Survival (FFS) at Two Years
Description: The two year rate of failure free survival (FFS) in study participants. This will include locoregional recurrence, and distant metastases. FFS is defined as absence of any failures (locoregional, distant metastasis, and death) during the time elapsed from the start of neoadjuvant chemotherapy to the date of documented failure events or radical cystectomy.
Time Frame: 2 Years
Population: as for outcome 1
Arm/Group | TURBT, NAC and Chemoradiation
Number analyzed (Participants) | 0

3. Secondary Outcome: Rate of Acute and Late Grade 2 or Higher Treatment-Related GU, GI and Hematologic Toxicity.
Description: The rate of acute and late grade 2 or higher (CTCAE v4.0) treatment-related genitourinary (GU), gastrointestinal (GI) and hematologic toxicity of bladder preservation in study participants.
Time Frame: Up to 2 years Post-Treatment
Population: as for outcome 1
Arm/Group | TURBT, NAC and Chemoradiation
Number analyzed (Participants) | 0

4. Secondary Outcome: Rate of Overall Survival in Study Participants
Description: Rate of Overall Survival in Study Participants. Overall survival (OS) is defined as the time elapsed from the start of neoadjuvant chemotherapy until death. Surviving patients (including patients lost to follow up) will be censored at the date of last contact.
Time Frame: Up to 3 years
Population: as for outcome 1
Arm/Group | TURBT, NAC and Chemoradiation
Number analyzed (Participants) | 0

5. Other Pre Specified Outcome: Evaluation of Known Predictive and Prognostics Biomarkers for Complete Response to Neoadjuvant Chemotherapy and Bladder Preservation.
Description: To evaluate known predictive and prognostic biomarkers for complete response to neoadjuvant chemotherapy and bladder preservation. Blood, urine and tumor tissue will be collected pre- and post-neoadjuvant chemotherapy, post-cystectomy or chemoradiation, and at any time point of distant metastases.
Time Frame: Up to 1 year Post-Treatment, About 2 years
Population: as for outcome 1
Arm/Group | TURBT, NAC and Chemoradiation
Number analyzed (Participants) | 0

6. Other Pre Specified Outcome: Identification of New Predictive and Prognostic Biomarkers for Response to Neoadjuvant Chemotherapy, and Bladder Preservation.
Description: To perform exploratory molecular analysis to identify new predictive and prognostic biomarkers for response to neoadjuvant chemotherapy, and bladder preservation. Blood, urine and tumor tissue for muscle invasive bladder cancer. Blood, urine and tumor tissue will be collected pre and post-neoadjuvant chemotherapy, post-cystectomy or chemoradiation, and at any time point of distant metastases.
Time Frame: Up to 1 year Post-Treatment, About 2 years
Population: as for outcome 1
Arm/Group | TURBT, NAC and Chemoradiation
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 2 years Post-Treatment
Arm/Group | TURBT, NAC and Chemoradiation
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TURBT, NAC and Chemoradiation (N=1)
Bloating (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 1 (1)
White blood cell decreased (Investigations) | 1 (3)
Platelet count decreased (Investigations) | 1 (1)
Mucositis/stomatitis (functional/symptomatic) (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
A minimum of 35 evaluable participants were required for the analysis of data for the study outcome measures. Fewer than the minimum number of participants required were enrolled therefore data were not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-07-15): https://cdn.clinicaltrials.gov/large-docs/90/NCT02145390/Prot_SAP_000.pdf